CLINICAL TRIAL: NCT05217524
Title: Evaluation of the Accuracy of a Novel Smartwatch Bioimpedance Device for Assessment of Body Composition
Brief Title: Samsung Galaxy Watch Body Composition Study
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Steven Heymsfield, Professor, Pennington Biomedical Research Center
Other Study IDs: PenningtonBRC
Record Dates: First submitted 2022-01-04; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pennington and Univ. of Hawaii cohorts: Same protocol but two different sites.
  Interventions: Device: Galaxy BIA watch
- Pennington: Primarily non-Hispanic (NH) White and NH Black at PBRC and more Asian and Native Hawaii or Pacific Islander (NHOPI) at Hawaii.
  Interventions: Device: Galaxy BIA watch

INTERVENTIONS:
Device: Galaxy BIA watch — Digital multifunction watch

SUMMARY:
The aim of this study is to acquire impedance measurements of the adult human body with a novel bioimpedance device housed inside a watch case and to compare derived estimates of body composition measured by dual-energy x-ray absorptiometry (DXA) and other bioimpedance analysis (BIA) systems.

DETAILED DESCRIPTION:
Aims:

The study hypothesis will be tested as follows. Each subject will complete novel BIA, DXA, anthropometric, and other BIA studies at PBRC and the University of Hawaii Cancer Center. The acquired data will then be used to accomplish the specific aims:

1. Identify the associations of body composition acquired by the novel BIA devices with those estimated by DXA and other BIA systems.
2. Describe the precision and accuracy of the novel BIA-derived body composition estimates.

Subjects and Design:

We will recruit a stratified sample of 100 participants recruited from the Baton Rouge metropolitan area for this study over a span of 6 months. Participants will be further subdivided into cohorts based on gender, age, and BMI.

The participants will be community dwelling and have no life-threatening conditions or diseases that would alter their body composition from what is typical for their age, sex, ethnicity, and BMI. Overall, participants must be ambulatory, able to withstand lying flat on the DXA table for up to 10 minutes, stand without aid for 2 minutes, weigh less than 440 lbs and be of generally good health.

Each subject enrolled in the study will have body weight, height, vital signs, urine testing (women of child bearing potential) and circumferences taken on the study visit day. Immediately after these measurements are completed, each subject will undergo a whole body DXA scan, and BIA measurements on the novel BIA and other BIA systems.

Recruitment and Screening Methods:

Subjects will be recruited through a web-based questionnaire, direct phone calls, media, and community outreach. Multiple forms of communication including paid advertisements such as print/social media/mass media etc. will be used to market the study and direct potential participants to the web site to complete the web screener application. In addition, the Recruitment Departments will participate in regional health events in which study information will be available to those interested in screening. A recruiter would then follow up with that participant to pre-screen them for the study.

The web screener / phone screening process will include the participant filling out basic health information, demographic information, as well as risk factors for metabolic conditions. A recruiter will follow up with all participants who are eligible via the web screener, phone in to the recruitment department, or show interest at a community event. If the subject is eligible, the recruiter will schedule their study visit.

A copy of the consent will be provided to subjects at the time of study visit. Subjects will be consented in a private room, and they can contact the investigators should any questions arise.

The subject will then fill out an electronic questionnaire regarding dietary history and physical activity.

Participants will be asked to arrive in gym-style clothing or clothing that is easily removable as they will be in form-fitting garments for all BIA, DXA, and tape measurements.

Study Endpoints:

The first aim is to recruit 100 participants stratified to cover the range of body sizes, BMI values, ethnicities, and ages for both sexes.

Measurements:

All subjects will have body circumferences, DXA, and BIA measurements. Note that times listed below include the subject moving from one lab to another.

Baseline evaluations: A series of body measurements will be taken by trained staff. These measurements include height, weight, and vital signs. The subject's BMI will be calculated from these measurements. An electronic questionnaire will be filled out (appended).

Body Composition Measurements

Circumferences Circumferences of the waist, hip, right upper arm and right thigh will be measured. The circumference measurements will be made by a trained clinical coordinator using a calibrated tape measure. We have an anthropometric training and validation program in place from earlier studies. These measurements will be made in about 20 minutes.

Novel BIA Body Composition will be measured using the novel BIA systems that takes under xx seconds per test. XX measurements will be made on each evaluation.

Dual-energy x-ray absorptiometry (DXA), (single measurement, about 20 minutes):

This scan measures the amount of bone, muscle, and fat, along with the mass of the head, arms, trunk, and legs. The scan will be performed using a whole-body scanner (Discovery System). The subject will be required to remove all metal-containing objects from the body and to lie down on the table. The subject will be carefully positioned on the table. A scanner emitting low energy X-rays and a detector will pass along the body. The subject will be asked to remain completely still while the scan is in progress. The scan will take approximately 10-15 minutes. Women of childbearing potential undergoing DXA will have a negative pregnancy test. DXA system operated according to manufacturer specifications.

Bioelectrical Impedance Analysis (BIA) (needs updating according to BIA systems used in the study) These tests will measure the amount of fat in the body. The subject will also be asked to lie down on an exam table and have electrodes attached to the hands and feet for BIA (InBody 570; Seoul, Korea): 2 consecutive measurements

This protocol presents minimal risks to the subjects, and adverse events or other problems are not anticipated. In the unlikely event that such events occur, Drs. Heymsfield and Shepherd are responsible for reporting serious, unanticipated and related adverse events or unanticipated problems involving risks to subjects or others to the IRB.

Timeframe:

The study will be completed over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* • • Being either male or female

  * Being from 18 to 80 years of age
  * Having a body weight of less than 440 pounds
  * Being willing to comply with the study procedures
  * Able climb 10 steps without difficulty and able to perform activities of daily living without difficulty (self-reported)

Exclusion Criteria• Being pregnant or attempting to become pregnant

* Having medical implants such as a pacemaker or metal joint replacements
* Having a body weight greater than 440 pounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy race/ethnically mixed adults
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
%body fat | 6 months
  Referenced against DXA

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marazzato F, McCarthy C, Field RH, Nguyen H, Nguyen T, Shepherd JA, Tinsley GM, Heymsfield SB. Advances in digital anthropometric body composition assessment: neural network algorithm prediction of appendicular lean mass. Eur J Clin Nutr. 2024 May;78(5):452-454. doi: 10.1038/s41430-023-01396-3. Epub 2023 Dec 23. PMID 38142263
- [Derived] McCarthy C, Tinsley GM, Yang S, Irving BA, Wong MC, Bennett JP, Shepherd JA, Heymsfield SB. Smartphone prediction of skeletal muscle mass: model development and validation in adults. Am J Clin Nutr. 2023 Apr;117(4):794-801. doi: 10.1016/j.ajcnut.2023.02.003. Epub 2023 Feb 8. PMID 36822238